CLINICAL TRIAL: NCT07310576
Title: Health Diet Education on Nutrition Literacy and Behavior
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: En-Chi Chiu (Other)
Collaborators: Taiwan Adventist Hospital (Other)
Responsible Party: Sponsor-Investigator, En-Chi Chiu, Associate Professor, National Taipei University of Nursing and Health Sciences
Organization: National Taipei University of Nursing and Health Sciences (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2025E09
Record Dates: First submitted 2025-12-16; First posted 2025-12-30 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Nutrition Status
Keywords: nutrition knowledge; dietary

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hospital staff (Experimental): Healthy diet interactive challenge program
  Interventions: Other: Nutritional knowledge
- Volunteer (Experimental): Senior nutrition and wellness course
  Interventions: Other: Nutritional knowledge

INTERVENTIONS:
Other: Nutritional knowledge — Healthy diet interactive challenge program: An engaging, game-based nutrition education activity designed to enhance participants' healthy eating knowledge and motivation through interactive challenges and practical dietary tasks.
  Senior nutrition and wellness course: A structured educational program for older adults focusing on balanced nutrition, healthy lifestyle habits, and practical strategies to promote overall well-being

SUMMARY:
This study was to investigate the effects of a health diet education program on improving nutrition knowledge, satisfaction, and dietary behavior among hospital staffs and volunteers.

DETAILED DESCRIPTION:
There were two groups: hospital staffs and volunteers.

ELIGIBILITY:
Inclusion Criteria:

* being willing to attend the program and complete the questionnaires
* providing inform consent to the use of their data for research analysis

Exclusion Criteria:

* Unable to complete the questionnaire (e.g., dementia, impaired consciousness, or severe visual impairment)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2025-09-10 (Actual); Primary Completion 2025-11-10 (Actual); Study Completion 2025-11-10 (Actual)

PRIMARY OUTCOMES:
Nutrition Knowledge questionnaire | Baseline to 2 months
  A self-administered survey designed to assess participants' understanding of healthy eating. The range of score was 1-6. A higher score indicated a greater level of knowledge about healthy eating.
Satisfaction and Behavioral Change Intention questionnaire | Baseline to 2 months
  A self-administered survey designed to assess participants' satisfaction with the educational program and intentions to adopt healthier dietary behaviors. The range of scores was 9-50, with higher scores indicating greater satisfaction and stronger intentions to adopt healthier dietary behaviors.

CONTACTS AND LOCATIONS:
Overall Officials: Shu-Chi Lin, MS, Principal Investigator — Taiwan Adventist Hospital
Locations (1):
- Taiwan Adventist Hospital, Taipei, Songshan District, Taiwan